CLINICAL TRIAL: NCT02251574
Title: Effect of a Very Low Calorie and Low Calorie Diet on Moderate to Severe Obstructive Sleep Apnea in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001418
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Caloric Restriction; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Calorie Diet (Experimental): Participants will take part in an experimental weight management program involving a low calorie diet (LCD), about 1200-1500 calories per day.
  Interventions: Other: Low Calorie Diet
- Very Low Calorie Diet (Experimental): Participants will take part in an experimental weight management program involving a low calorie diet (LCD), about 520-800 calories per day.
  Interventions: Other: Very Low Calorie Diet
- Standard Care (Active Comparator): Participants will receive normal care.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Low Calorie Diet — Weight management program designed around a low calorie diet.
  Arms: Low Calorie Diet
Other: Very Low Calorie Diet — Weight management program designed around a very low calorie diet.
  Arms: Very Low Calorie Diet
Other: Standard Care — Care provided that would normally be given to people meeting eligibility criteria for this study.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to test the effectiveness of two different weight loss diets on obstructive sleep apnea (OSA) severity.

DETAILED DESCRIPTION:
Sleep apnea is a sleep disorder in which breathing repeatedly stops and starts during sleep. The most common type is obstructive sleep apnea (OSA), which occurs when the muscles in your throat relax and block your airway during sleep. The most noticeable sign of OSA is snoring. OSA is a risk factor for other chronic conditions like type 2 diabetes, cardiovascular disease, and high blood pressure.

Although anyone can develop OSA, it commonly affects people who are obese. The more someone weighs, the more likely the OSA is to be severe. Weight loss is typically recommended for overweight individuals to help improve OSA. However, not enough research has been done for doctors to be able make specific recommendations to their patients.

ELIGIBILITY:
Inclusion Criteria:

* AHI score of ≥ 5
* Body mass index (BMI) between 30 to 49.9 kg/m2

Exclusion Criteria:

* Report serious medical risk such as insulin-dependent diabetes, active cancer, recent cardiac event
* Currently or planning to become pregnant during the next 9 months
* Not weight stable (-4.6 kg) for 3 mos. prior to intake
* Report current participation in a weight reduction program involving diet or PA
* Unwilling to be randomized to 1 of 3 study groups
* Report symptomology of an eating disorder as determined by the Eating Attitudes Test
* Unable to participate in moderate intensity physical activity

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI) | Change from Baseline to Month 3
  The AHI measures sleep apnea severity and represents the number of apnea and hypopnea events per hour.

SECONDARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI) | Change from Baseline to Month 9
  The AHI measures sleep apnea severity and represents the number of apnea and hypopnea events per hour.
Change in metabolic syndrome (MetS) risk factors | Change from Baseline to Month 3 and Month 9
  Risk factors to be measured include waist circumference, triglycerides, HDL-cholesterol, blood pressure, fasting glucose
Change in Quality of Life | Change from Baseline to Month 3 and Month 9
  Participants will complete the Calgary Sleep Apnea Quality of Life Index (SAQLI) that will assess participants response to the intervention/treatment.
Change in Daytime Sleepiness | Change from Baseline to Month 3 and Month 9
  Researchers will administer Epworth Sleepiness Scale. Results will be used to calculate daytime sleepiness changes for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine Goetz, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States